CLINICAL TRIAL: NCT01465841
Title: ACE: An Aneurysm Coiling Efficiency Study of the Penumbra Coil 400 System
Brief Title: Study of the Penumbra Coil 400 System to Treat Aneurysm
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 4492; CLP 4492 (Other: Penumbra Inc)
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Intracranial Aneurysms; Peripheral Aneurysms
Keywords: intracranial aneurysms; Peripheral aneurysms; acute treatment; PC 400 System; packing density
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Embolization with the PC 400 coils (Experimental)
  Interventions: Device: PC 400 coils (Penumbra )

INTERVENTIONS:
Device: PC 400 coils (Penumbra ) — The Penumbra Embolization Coil is indicated for the endovascular embolization of aneurysms. The Embolization Coil functions to selectively embolize aneurysms by packing a sufficient quantity of soft platinum coils to achieve occlusion. The Coil Implant is constructed of 92% Platinum and 8% Tungsten round wire with a diameter approximately 0.0015in ± 0.0001in. The maximum primary diameter is 0.022in and the coil implant will have a semi-spherical atraumatic distal tip.

SUMMARY:
This is a prospective, multi-center study of patients with intracranial or peripheral aneurysms who are treated by the PC 400 System. The primary objective is to gather post market data on the Penumbra Coil 400 (PC 400) System in the acute treatment of intracranial and peripheral aneurysms. Approximately 2,000 patients with intracranial or peripheral aneurysms treated by the PC 400 System at up to 100 centers will be enrolled. Data for each patient are collected up to discharge or 3 days post-procedure, whichever occurs sooner. Long term follow-up to one year will be conducted in accordance to the standard of care at each participating hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in this study must be those treated according to the cleared indication for the PC 400 System which is for the endovascular embolization of:

* Intracranial aneurysms
* Other neurovascular abnormalities such as arteriovenous malformations and arteriovenous fistulae
* Arterial and venous embolizations in the peripheral vasculature

Exclusion Criteria:

* Patients in whom endovascular embolization therapies other than Penumbra Coils are used will be excluded from this study. However, adjunctive use of balloon and stent are acceptable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2011-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siu P Sit, PhD, Study Director — Penumbra Inc.
Locations (6):
- United States (6):
  - Hoag Hospital, Newport Beach, California
  - Rush University Medical Center, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - State University of New York Upstate Medical Center, Syracuse, New York
  - Fort Sanders Medical Center, Knoxville, Tennessee
  - The Methodist Hospital Research Institute, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Embolization With the PC 400 Coils
Started | 517
Completed | 449
Not Completed | 68

BASELINE CHARACTERISTICS:
Arm/Group | Embolization With the PC 400 Coils
Number analyzed (Participants) | 517
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (14.4)
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 365
  Male | 152
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Packing Density With the Number of Coils Implanted
Description: The data will be captured at the end of the coiling procedure which is standard for aneurysm studies.
Time Frame: At immediate post-procedure
Measure: Mean (Standard Deviation); unit: percentage of aneurysm volume
Arm/Group | Embolization With the PC 400 Coils
Number analyzed (Participants) | 416
percentage of aneurysm volume | 37.9 (15.9)

2. Primary Outcome: Time of Fluoroscopic Exposure
Description: The total time of fluoroscopic exposure will be captured from the initial recording of the road map to the final angiogram after completion of the coiling procedure.
Time Frame: At immediate post-procedure
Population: The analysis population includes all intent-to-treat population. Procedural fluoroscopy time was available for 533 subjects.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: lesions
Arm/Group | Embolization With the PC 400 Coils
Number analyzed (Participants) | 517
Number analyzed (lesions) | 533
minutes | 38.2 (28.9)

3. Primary Outcome: Procedural Device-related Serious Adverse Events
Description: Procedural on-the-table serious adverse events will be captured and recorded at the end of the procedure. The duration of the procedure can be variable, depending on the time to access the target lesion and the time to complete the coiling procedure.
Time Frame: At immediate post-procedure
Measure: Number; unit: events
Arm/Group | Embolization With the PC 400 Coils
Number analyzed (Participants) | 517
events | 12

4. Secondary Outcome: Acute Occlusion of the Aneurysm Sac
Description: Measured using Raymond Roy classification where grading ranges from I to III and higher values represent a worse outcome.
Time Frame: At immediate post-procedure
Measure: Number; unit: participants
Arm/Group | Embolization With the PC 400 Coils
Number analyzed (Participants) | 465
participants
  Raymond-Roy Occlusion Class I | 214
  Raymond-Roy Occlusion Class II | 136
  Raymond-Roy Occlusion Class III | 115

5. Secondary Outcome: Intracranial Hemorrhage
Time Frame: At discharge or 3 days post-procedure
Measure: Number; unit: events
Arm/Group | Embolization With the PC 400 Coils
Number analyzed (Participants) | 517
events | 4

ADVERSE EVENTS:
Time Frame: up to 1 year in accordance to the standard of care at participating hospitals
Arm/Group | Embolization With the PC 400 Coils
All-Cause Mortality (participants affected / at risk) | 32/517
Serious Adverse Events (participants affected / at risk) | 126/517
Other Adverse Events (participants affected / at risk) | 284/517
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Embolization With the PC 400 Coils (N=517)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3
Cardiac Disorders (Cardiac disorders) | 10
Congenital, familial, and genetic disorders (Congenital, familial and genetic disorders) | 1
Eye Disorders (Eye disorders) | 1
Gastrointestinal Disorders (Gastrointestinal disorders) | 15
General Disorders and Administration Site Conditions (General disorders) | 14
Hepatobiliary Disorders (Hepatobiliary disorders) | 3
Infections and Infestations (Infections and infestations) | 17
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 10
Investigations (Investigations) | 1
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 5
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 3
Neoplasms Benign, Malignant and Unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Nervous System Disorders (Nervous system disorders) | 63
Psychiatric Disorders (Psychiatric disorders) | 3
Renal and Urinary Disorders (Renal and urinary disorders) | 2
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 14
Surgical and Medical Procedures (Surgical and medical procedures) | 2
Vascular Disorders (Vascular disorders) | 20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Embolization With the PC 400 Coils (N=517)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 10
Cardiac Disorders (Cardiac disorders) | 22
Congenital, familial, and genetic disorders (Congenital, familial and genetic disorders) | 1
Ear and Labyrinth Disorders (Ear and labyrinth disorders) | 3
Endocrine Disorders (Endocrine disorders) | 1
Eye Disorders (Eye disorders) | 20
Gastrointestinal Disorders (Gastrointestinal disorders) | 47
General Disorders and Administration Site Conditions (General disorders) | 65
Hepatobiliary Disorders (Hepatobiliary disorders) | 4
Immune System Disorders (Immune system disorders) | 1
Infections and Infestations (Infections and infestations) | 43
Injury, Poisoning, and Procedural Complications (Injury, poisoning and procedural complications) | 26
Investigations (Investigations) | 13
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 21
Muskuloskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 18
Neoplasms Benign, Malignant, and Unspecified (inc cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Nervous System Disorders (Nervous system disorders) | 160
Psychiatric Disorders (Psychiatric disorders) | 22
Renal and Urinary Disorders (Renal and urinary disorders) | 12
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 30
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 8
Surgical and Medical Procedures (Surgical and medical procedures) | 4
Vascular Disorders (Vascular disorders) | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01465841/Prot_SAP_000.pdf